CLINICAL TRIAL: NCT01774435
Title: A Phase 1, Open-Label, Study in Stabilized Schizophrenic Patients to Evaluate the Pharmacokinetics of Risperidone and 9-Hydroxy (OH) Risperidone When Risperidone is Administered From a Polyurethane Implant
Brief Title: Study in Stabilized Schizophrenic Patients to Evaluate the Pharmacokinetics of Risperidone and 9-Hydroxy (OH)-Risperidone When Risperidone is Administered From a Polyurethane Implant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3342-102
Record Dates: First submitted 2013-01-07; First posted 2013-01-24 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic; Stable Schizophrenic
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EN3342 (Experimental): EN3342 (risperidone) subcutaneous implant
  Interventions: Drug: EN3342

INTERVENTIONS:
Drug: EN3342

SUMMARY:
This is an study evaluating the safety, tolerability, and PK of EN3342 in implantation durations of 6 months.

ELIGIBILITY:
Subject Inclusion Criteria

1. Subject (and/or a subject's authorized legal representative) has provided written informed consent
2. Subject has identified a caregiver or personal contact with whom the subject has significant contact with at least once per week
3. Subject is male or female of non-child bearing potential between 18 to 60 years of age inclusive
4. Subject has a diagnosis of schizophrenia according to DSM-IV criteria
5. Subject has a body mass index (BMI) ≥18.5 and ≤35.0 kg/m2
6. Subject is assessed to be symptomatically stable by the Investigator, with regard to his or her psychiatric condition
7. Subject is assessed by the Investigator to be symptomatically stable with regard to pre existing medical conditions as evidenced by medical history, clinically significant findings on physical examination, vital signs, clinical laboratory evaluations (hematology, serum chemistries, and urinalysis) or 12-lead electrocardiogram (ECG). Subjects may continue on their current medication regimen to control pre-existing medical and psychiatric (other than schizophrenia) conditions including the use of PRN medications.
8. Subject is currently stable on a 4-, 6-, or 8-mg oral dose of risperidone for 30 days prior to admission

Subject Exclusion Criteria

1. Known hypersensitivity or allergy to lidocaine or any local anesthetic agent of the amide type (local anesthetic used during implant and explant procedures)
2. Known sensitivity to polyurethane
3. Hospitalized or required acute crisis intervention for symptom exacerbation in the 30 days prior to admission as determined by the Investigator
4. Subject has a history of suicide attempt in the last year, or in the opinion of the investigator is currently at imminent risk of suicide
5. Reports or reveals a presence of clinically significant skin disorders (such as, but not limited to, skin cancer, psoriasis, eczema, or atopic dermatitis), evidence of recent sunburn, scar tissue, tattoo, open sore, body piercing or branding at the intended implantation site that would interfere with the implantation procedure or interfere with implant site assessments as determined by the Investigator
6. History of abnormal scar formation or family history of keloid formation
7. Have a positive screen for substances of abuse conducted at screening or had any history of abuse in the last six months as defined by DSM-IV criteria
8. Have impaired hepatic (ALT/AST >1.5 times higher than the upper limit of normal) or renal function (eGFR <50mL/min)
9. Previously defined hypersensitivity to risperidone
10. History of neuromalignant syndrome (NMS)
11. Electroconvulsive therapy within 6 months of admission
12. Treatment of coexisting medical conditions that require the introduction of cytochrome P450 2D6 inhibitors or inducers
13. Positive screen for Hepatitis B Surface Antigen (HBsAg), Hepatitis C Antibody (anti HCV), or human immunodeficiency virus (HIV) antibody and/or antigen
14. Participation in the treatment phase of a clinical study or receipt of an investigational drug within 30 days prior to study drug administration on Day 1; for investigational drugs with an elimination half-life greater than 15 days, this time period will be extended to 60 days
15. Prior participation in a EN3342 study
16. Involvement in the planning and/or conduct of the study (applies to both Endo staff or staff at the investigational site)
17. History of difficulty with phlebotomy procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
PK parameters (Cmax and AUC) for active moiety, 9-OH-risperidone and risperidone | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Litman, MD, Principal Investigator — CBH Health LLC
Locations (1):
- CRI Lifetree, Marlton, New Jersey, United States